CLINICAL TRIAL: NCT04093661
Title: Retrospective Analysis of Intraoperative Electroencephalography Characteristics in Children Under One Year of Age
Brief Title: Electroencephalogram Dynamics in Children <=1 Year During Anesthetic Procedures
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Claudia Spies, Head of the Department of Anesthesiology and Operative Intensive Care Medicine (CCM/CVK), Charite University, Berlin, Germany
Other Study IDs: Retro-Baby
Record Dates: First submitted 2019-09-16; First posted 2019-09-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Depth of Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children below 1 year: Children <= 1 year for elective surgery

SUMMARY:
As part of the clinical routine of the Department of Anesthesiology and Operative Intensive Care Medicine (CCM/CVK), Charité - Universitätsmedizin Berlin at Campus Virchow-Klinikum intraoperative electroencephalography data and clinical routine data are recorded and evaluated in surgical children (<=1 year).

ELIGIBILITY:
Inclusion Criteria:

• Children <= 1 year undergoing surgery procedure

Exclusion Criteria:

* Incomplete patient record documentation
* Pre-existing neurological/psychological conditions

Ages: 1 Month to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children <= 1 year undergoing surgery procedure with Electroencephalography Monitoring.
Sampling Method: Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2019-11-29 (Actual); Study Completion 2019-11-29 (Actual)

PRIMARY OUTCOMES:
Electroencephalography monitoring changes | 06/2017 - 06/2019
  The primary objective of this study performed according to an observational post-ad-hoc design measures the perioperative EEG overall power signature. Approximately 150 children admitted from 06/2017 to 06/2019 to the Charité will be enrolled in the study. They are followed up until their discharge from the recovery room.

SECONDARY OUTCOMES:
Anesthetic depth | 06/2017 - 06/2019
  Anesthetic stage is related to typical time points during an anesthetic procedure - as "loss of consciousness", "intubation", "stable anesthesia", "extubation", "regain of consciousness". Approximately 150 children admitted from 06/2017 to 06/2019 to the Charite will be enrolled in the study. They are followed up until their discharge from the recovery room.
Medication | 06/2017 - 06/2019
  Medication data are captured from the patient sheets. Approximately 150 children admitted from 06/2017 to 06/2019 to the Charite will be enrolled in the study. They are followed up until their discharge from the recovery room.
Emergence Delirium | 06/2017 - 06/2019
  Delirium is captured form the PAED Score data in the patient records. Approximately 150 children admitted from 06/2017 to 06/2019 to the Charite will be enrolled in the study. They are followed up until their discharge from the recovery room.
Pain | 06/2017 - 06/2019
  Pain scores are captured form the patient records. Approximately 150 children admitted from 06/2017 to 06/2019 to the Charite will be enrolled in the study. They are followed up until their discharge from the recovery room.

OTHER OUTCOMES:
Duration of anesthesia | 06/2017 - 06/2019
  Duration of anesthesia is captured from the patient records and measured until the end of surgery. Approximately 150 children admitted from 06/2017 to 06/2019 to the Charite will be enrolled in the study.
Type of surgery | 06/2017 - 06/2019
  Type of surgery is captured from the patient records. Approximately 150 children admitted from 06/2017 to 06/2019 to the Charite will be enrolled in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, MD, Prof., Study Director — Department of Anesthesiology and Operative Intensive Care Medicine, Campus Charité Mitte and Campus Virchow-Klinikum, Charité - Universitätsmedizin Berlin
Locations (1):
- Department of Anesthesiology and Operative Intensive Care Medicine (CCM/CVK), Charité - Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No